CLINICAL TRIAL: NCT01279616
Title: A Pilot Study of an Immunosuppressive and Myeloablative Preparative Regimen for Allogeneic Unrelated Donor Hematopoietic Stem Cell Transplantation (HSCT) for Severe Sickle Cell Disease
Brief Title: A Reduced Toxicity Allogeneic Unrelated Donor Stem Cell Transplantation (SCT) for Severe Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI moving to a different institution.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-00383
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell; stem cell transplant
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — fludarabine phosphate; Rituximab; Busulfan; thymoglobulin; Cyclophosphamide; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic Stem Cell Transplant (Experimental): Stem cell infusion on Day 0.
  Interventions: Drug: Fludarabine monophosphate; Drug: Rituximab; Drug: Busulfan; Drug: ATG; Drug: Cyclophosphamide; Drug: Mycophenolate mofetil; Drug: Tacrolimus

INTERVENTIONS:
Drug: Fludarabine monophosphate — 180 mg/m2 over 6 days.
Drug: Rituximab — 375 mg/m2 on day -13 and day -3
  Other Names: Rituxan
Drug: Busulfan — AUC 1000-1200 microM.mt
  Other Names: busulfex
Drug: ATG — 2.5 mg/kg for 3 days
  Other Names: Thymoglobulin
Drug: Cyclophosphamide — 50 mg/kg on day +3
  Other Names: Cytoxan
Drug: Mycophenolate mofetil — 15 mg/kg q 8 hours
  Other Names: MMF, Cell-cept.
Drug: Tacrolimus — 0.03 mg/kg /d
  Other Names: FK-506

SUMMARY:
Majority of patients who are eligible for allogeneic HSCT for cure of severe sickle cell disease lack a matched family donor. This study aims for cure of sickle cell disease by performing unrelated donor (outside family) allogeneic HSCT. Donors or unrelated cord blood units will be selected from the NMDP database. It is designed to estimate the safety of a novel reduced toxicity, yet an immunosuppressive and myeloablative preparative regimen. This is meant for patients <21 years old who have severe complications from sickle cell and do not have matched sibling donors in the family to undergo stem cell transplant. Patients will undergo transplant using unrelated donor stem cells after receiving the protocol therapy. They will be followed for 1 year to monitor for engraftment of donor cells and complications like graft versus host disease (GVHD), infections and death.

DETAILED DESCRIPTION:
The primary goal of this pilot study is to determine the safety and feasibility of the preparative regimen for HSCT using a novel reduced toxicity regimen for stem cell transplant with unrelated donors. Analysis will be geared to confirm if the study regimen, followed by an appropriately HLA-matched unrelated donor (MUD)or unrelated cord blood HSCT, can lead to durable donor engraftment with reasonable toxicity, inhibiting sickle erythropoiesis and limiting disease related organ toxicity in patients who are at high risk for morbidity and mortality associated with sickle cell disease (SCD).

ELIGIBILITY:
Inclusion Criteria:

Patients must have sickle cell disease (genotype Hb SS or Sß° thalassemia), AND must have 1 or more of the following clinical complications related to Sickle cell disease:

1. A clinically significant neurologic event (stroke) or any neurologic defect lasting >24 hours, that is accompanied by an infarct on cerebral MRI.
2. Minimum of two episodes of acute chest syndrome (defined as new pulmonary alveolar consolidation involving at least 1 complete lung segment associated with acute symptoms including fever, chest pain, tachypnea, wheezing or cough) despite adequate supportive care measures (example: asthma therapy, hydroxyurea).
3. History of severe pain episodes defined as 3 or more severe pain events per year in the 2 years prior to enrollment despite adequate supportive care measures and hydroxyurea trial (i.e. Hydroxyurea non-responders). Pain may occur in typical sites associated with vaso-occlusive painful events and cannot be explained by causes other than vaso-occlusion mediated by sickle cell disease.
4. Recurrent priapism.
5. Osteo-necrosis of multiple joints
6. Evidence of Pulmonary Hypertension as evidenced by Tricuspid Regurgitation jet velocity (TRV) > 2.5 m/s on Echocardiogram.
7. Red cell allo-immunization (≥ 2 antibodies) during long term transfusion therapy.

Exclusion Criteria:

1. Invasive bacterial, viral or fungal infections within 1 month prior to starting conditioning therapy.
2. Female patients who are Pregnant (Beta HCG +) or breastfeeding.
3. HIV positive patients.
4. Patients with HLA-matched related family donors are not eligible for this study.
5. Prior myeloablative allogeneic HCT.
6. Patients on chronic transfusion therapy for ≥ 1 year with evidence of cirrhosis of liver on biopsy
7. Any significant concurrent disease, illness, severe cognitive delay or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Soni, MD, Study Chair — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Stem Cell Transplant: Drug: Fludarabine monophosphate 180 mg/m2 over 6 days.
  Drug: Rituximab 375 mg/m2 on day -13 and day -3 Other Names: •Rituxan
  Drug: Busulfan AUC 1000-1200 microM.mt Other Names: •busulfex
  Drug: ATG 2.5 mg/kg for 3 days Other Names: •Thymoglobulin
  Drug: Cyclophosphamide 50 mg/kg on day +3 Other Names: •Cytoxan
  Drug: Mycophenolate mofetil 15 mg/kg q 8 hours Other Names: •MMF, Cell-cept.
  Drug: Tacrolimus 0.03 mg/kg /d Other Names: •FK-506
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplant
Started | 8
Completed | 1
Not Completed | 7
Not completed — donor could not be located | 5
Not completed — no signs of sickle cell disease | 2

BASELINE CHARACTERISTICS:
Population: No baseline data are available for this study as the study was terminated. The PI has left the institution and cannot be contacted.
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]
Study-Specific Measure

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Event-free survival
Time Frame: 1 year
Population: The study was terminated and the PI has left the institution. Efforts were made to contact the PI but unsuccessful. No outcome measure data is available for the study.
Groups:
- HSCT Transplant: HSCT transplant
Arm/Group | HSCT Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From enrollment of first participation to study termination.
Description: The study was terminated and the PI has left the institution. The only available information is in respect to the serious adverse events.
Groups:
- No Arm Analyzed: N/A: No outcome date are available for this study as the study was terminated. The PI has left the institution and cannot be contacted.
Arm/Group | No Arm Analyzed: N/A
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No outcome data are available for this study as the study was terminated. The PI has left the institution and cannot be contacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No Outcome data are available for this study as the study was terminated. The PI has left the institution and cannot be contacted.